CLINICAL TRIAL: NCT03894111
Title: Prognostic Effect of Neutrophil \ Lymphocyte Ratio, Lactate Level and Apache 2 Score on Mortality in Intensive Care Trauma Patients at First Hospitalizations
Brief Title: ICU Mortality Predictors of Trauma Patients
Status: Completed | Type: Observational
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, bülent atik, asistant prof, Balikesir University
Other Study IDs: 2019/32
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: İntensive Care Unit
Keywords: trauma, mortality
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- living patients: living patients in intersivecare unit about 28 days
  Interventions: Other: decesased patients
- deceased patients: deceased patients in intersivecare unit about 28 days
  Interventions: Other: decesased patients

INTERVENTIONS:
Other: decesased patients — mortality ratio

SUMMARY:
In this study, the data of the patients who were hospitalized due to trauma in intensive care unit (ICU) were examined in their first development. The mortality rate and the factors affecting mortality in these patients were determined

DETAILED DESCRIPTION:
In this study, 107 trauma patients were examined. Patients were divided into two groups according to ICU results: survivors (Group 1) and deceased patients (Group2). Patients were rated in terms of age, Neutrophil lymphocyte ratio (NLR) , mean platelet volüme (MPV), lactat value, intensive care unit stay, APACHE 2 soring systems. Mortality rate and the factors affecting this rate were examined.

83 of the patients were male (77.58%) and 24 were female (22.42%). The mean age was 46 years. The mean value of lactate level was 3.25. MPV mean value was 10.34. NLR mean value was 8.23 and Apache 2 score mean value was 22.8. The average length of stay in hospital was 11.33 days. When the intergroup mortality was evaluated in terms of the relationship between continuous variables, there was a statistically significant difference in apache 2 score. No statistically significant difference was found between age, lactate, MPV, NRL and length of hospital stay.

NRL, MPV, Lactate levels were not suitable for evaluation of trauma patients as a early prognostic factor in the first day ICU admission. The investigators think that the use of trauma scoring systems such as apache 2 related to mortality during first hospitalization in ICU is more appropriate.

ELIGIBILITY:
Inclusion Criteria:

* trauvma patients

Exclusion Criteria:

* systemic inflammatory diseases
* cancer
* renal failure
* cardiac failure
* serebro vascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all trauvma patients in one year
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
mortallty | 28 days
  mortallty ratio

CONTACTS AND LOCATIONS:
Overall Officials: bülent atik, md, Principal Investigator — Netherlands: Ministry of Health, Welfare and Sports
Locations (1):
- Balikesir City Hospital, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zahorec R. Ratio of neutrophil to lymphocyte counts--rapid and simple parameter of systemic inflammation and stress in critically ill. Bratisl Lek Listy. 2001;102(1):5-14. English, Slovak. PMID 11723675
- [Background] Chen W, Yang J, Li B, Peng G, Li T, Li L, Wang S. Neutrophil to Lymphocyte Ratio as a Novel Predictor of Outcome in Patients With Severe Traumatic Brain Injury. J Head Trauma Rehabil. 2018 Jan/Feb;33(1):E53-E59. doi: 10.1097/HTR.0000000000000320. PMID 28520670
- [Result] Dilektasli E, Inaba K, Haltmeier T, Wong MD, Clark D, Benjamin ER, Lam L, Demetriades D. The prognostic value of neutrophil-to-lymphocyte ratio on mortality in critically ill trauma patients. J Trauma Acute Care Surg. 2016 Nov;81(5):882-888. doi: 10.1097/TA.0000000000000980. PMID 26825931